CLINICAL TRIAL: NCT02872883
Title: "Active vs Expectant Management and Routine vs Only-when-necessary Vaginal Examinations During Labour for Prelabour Rupture of Membranes at Term, a Pilot RCT Study"
Brief Title: A Pilot RCT on the Management of Term Prelabour Rupture of Membranes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Central Lancashire (Other)
Collaborators: Lancashire Care NHS Foundation Trust (Network)
Responsible Party: Principal Investigator, Lucia Ramirez-Montesinos, Miss, University of Central Lancashire
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: STEMH-503; U1111-1185-3426 (Other: (Universal Trial Number)The World Health Organisation)
Record Dates: First submitted 2016-07-14; First posted 2016-08-19 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Prelabour Rupture of Membranes at Term
Keywords: Prelabour rupture of membranes; term pregnancy; management; vaginal examination; induction of labour; expectant management
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Expectant management and minimal vaginal examinations (Experimental): Expectant management up to approximately 96hours and vaginal examinations only when necessary during active labour
  Interventions: Procedure: Expectant management; Procedure: Minimal Vaginal examinations (only when necessary)
- Expectant management and routine vaginal examinations (Experimental): Expectant management up to approximately 96hours and routine vaginal examinations during active labour
  Interventions: Procedure: Expectant management; Procedure: Routine vaginal examinations
- Active management and minimal vaginal examinations (Experimental): Induction of labour at approximately 24hours and vaginal examinations only when necessary during active labour
  Interventions: Procedure: Minimal Vaginal examinations (only when necessary); Procedure: Active management
- Active management and routine vaginal examinations (Active Comparator): Induction of labour at approximately 24hours and routine vaginal examinations
  Interventions: Procedure: Active management; Procedure: Routine vaginal examinations

INTERVENTIONS:
Procedure: Expectant management
  Arms: Expectant management and minimal vaginal examinations; Expectant management and routine vaginal examinations
Procedure: Minimal Vaginal examinations (only when necessary)
  Arms: Active management and minimal vaginal examinations; Expectant management and minimal vaginal examinations
Procedure: Active management
  Arms: Active management and minimal vaginal examinations; Active management and routine vaginal examinations
Procedure: Routine vaginal examinations
  Arms: Active management and routine vaginal examinations; Expectant management and routine vaginal examinations

SUMMARY:
This is a pilot study that will eventually result in a main randomised controlled trial that will look at what management is associated with a higher rate of normal birth and a lower rate of chorioamnionitis (maternal infection) when women break their waters but labour does not start. Spontaneous rupture of the membranes (when the waters break) at term (37-42 weeks gestation) is a physiological event that happens during labour. However, according to Gunn et al. (1970) in 8-10 % of the cases the membranes rupture before labour starts. The time between the rupture and the onset of labour is called latent phase and time wise is variable.

Studies have showed no statistically significant differences in terms of neonatal infection or chorioamnionitis when the investigators induce labour with prostaglandins compared to when labour starts spontaneously (Hannah et al 1996). Seaward et al. (1997) noted a number of confounding factors that might relate to the incidence of chorioamnionitis (maternal infection), the strongest predictor was having more than 8 vaginal examinations since the rupture of membranes and before delivery which was a stronger predictor than the duration of the latent phase. It is thought that by reducing the number of internal examinations, chorioamnionitis may be reduced, and hence neonatal infection may also be reduced. The main RCT will compare clinical outcomes and maternal satisfaction when women consent to be randomized to four groups: (1) Active management and routine internal examinations during labour, (2) Active management and reduced internal examinations, (3) Expectant management and routine internal examinations, (4) Expectant management and reduced internal examinations.

This application seeks ethics approval for the pilot phase to ensure that a definitive study can be undertaken appropriately. It is important to test that all the components work well individually and as a whole, to estimate sample size and ultimately to test the integrity of the research protocol before embarking on the main trial.

ELIGIBILITY:
Inclusion Criteria:

* Prelabour rupture of membranes (confirmed)
* Term pregnancy - from 37+0 till 41+2 weeks gestation (both inclusive)
* Normal/Low risk pregnancy
* Singleton, cephalic pregnancy
* No known current infectious diseases
* Aged 18-45 years old
* Understands English and is able to read and write in English
* Agree for their placentas to be sent to histology if clinical signs of infection
* Not taking part in other clinical research at present
* Consent to take part

Exclusion criteria:

* Pregnancy of 36+6 or less or 41+3 or more weeks gestation
* Breech or oblique presentation
* Twin or multiple pregnancy
* Previous caesarean section
* Meconium stained liquor
* Pre-eclampsia
* Diabetes
* Known to be colonised by Group B streptococcus
* Current infections: HIV, Hepatitis B, Herpes
* Doesn't give consent for the placenta to be sent to histology if clinical signs of infection
* Not able to understand, read or write in English
* Currently taking part in other clinical research

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-10 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of eligible women who agree to take part in the study | 12 months during pilot stage

SECONDARY OUTCOMES:
Percentage of participants who stay in the allocation arm | 12 months during pilot stage
Percentage of participants who find the interventions acceptable | The questionnaire will be completed by the participants between 4-8 weeks after giving birth
  Acceptability of the interventions to participants as measured by the study questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Ramirez-Montesinos, MSc BSc, Principal Investigator — University of Central Lancashire; Soo Downe, PhD MSc BSc, Study Director — University of Central Lancashire
Locations (1):
- Lancashire Teaching Hospitals NHS Trust, Preston, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No